CLINICAL TRIAL: NCT05804136
Title: A Prospective Randomized Controlled Trial Comparing Duramesh™ With Polydioxanone Suture for Laparotomy Closure
Brief Title: Duramesh™ vs Polydioxanone Suture for Laparotomy Closure
Acronym: MOMENTUM RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOMENTUM RCT ONZ-2022-0507
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Laparotomy Closure After Abdominal Surgery

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, academic, prospective, randomized-controlled, interventional, monocenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Duramesh (Other): Laparotomy closure is associated with the occurrence of Surgical Site Events (SSEs) such as wound dehiscence and incisional hernias. Abdominal wall closure can also cause pain and discomfort, or can lead to intestinal obstruction.
  Standard sutures can cut through otherwise intact tissue due to the presence of a sharp leading edge leading to repair failure. Meshes distribute forces and allow for tissue ingrowth. Duramesh combines the desirable principles of a mesh repair with the placement precision of a suture. It is the world's first device that both approximates tissue and allows ingrowth for a strong early repair.
  Consequently, the expected clinical benefit is the reduced occurrence of Surgical Site Events such as incisional hernias. Additional benefits may include reduced pain and improved quality of life due to durable closure of the abdominal wall with Duramesh. This will be evaluated in this randomized study.
  Size 1 Duramesh is used in this RCT. Duramesh is CE-marked.
  Interventions: Device: Duramesh
- Standard suture (Other): 2-0, 0, or Number 1 polydioxanone suture (PDS) is used as comparator.
  Interventions: Device: Polydioxanone suture

INTERVENTIONS:
Device: Duramesh — Laparotomy closure with Duramesh
  Arms: Duramesh
Device: Polydioxanone suture — Laparotomy closure with standard PDS
  Arms: Standard suture

SUMMARY:
This study is intended to demonstrate the non-inferiority of a Duramesh closure as compared to a polydioxanone closure for early surgical site events (SSE) (< 1 month), and Duramesh superiority to polydioxanone for the development of incisional hernia by 1 year for a laparotomy closure.

DETAILED DESCRIPTION:
This clinical investigation is designed to compare laparotomy closure with Duramesh to closure using PDS. The primary outcome is SSE that occurs within 1 month after surgery. Secondary outcomes that will be studied include device performance and technical success of the index-procedure, hernia occurrence/recurrence noted at 12 months after surgery, SSE and re-interventions that occur within 12 months of surgery, pain, implant palpability/sensation, surgeon and patient satisfaction, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Abdominal laparotomy 5 cm in length or greater, either midline or non-midline
* Isolated ostomy site takedown with or without parastomal hernia
* Patient accepts participation and gives informed consent
* Patient and investigator signed and dated the informed consent form prior to the index-procedure

Exclusion Criteria:

* Pregnancy
* Presence of clinically recognized hernia at laparotomy site (parastomal hernia noted at time of ostomy site takedown is not an exclusion criterion. Subclinical incidental small hernia < 1 cm in greatest dimension found at the time of a laparotomy is not an automatic exclusion criterion)
* Prior hernia repair at laparotomy site
* Use of planar mesh in addition to sutures for closure
* CDC IV dirty or infected wound that causes the surgeon to leave the abdominal wall or skin incision open
* Life expectancy less than 1 year
* Patient is unable / unwilling to provide informed consent
* Patient is unable to comply with the protocol or proposed follow-up visits
* Patient is enrolled in another abdominal wall study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is SSE that occurs within 1 month after surgery. | 1 month
  This study is intended to demonstrate the non-inferiority of a Duramesh closure as compared to a polydioxanone closure for early surgical site events (SSE) (< 1 month).
  SSE include: Seroma, Hematoma, Soft tissue breakdown, Fascial dehiscence, Cellulitis, Suture granuloma, Chronic draining sinus, Enterocutaneous fistula, Superficial, deep and organ/space infections, Other

SECONDARY OUTCOMES:
SSE within the first 12 months after repair. | 12 months
  SSE include: Surgical incision wound (this does NOT include a less than 5 mm scar-related superficial wound due to scar instability), Chronic draining sinus, Enterocutaneous fistula, Persistent seroma or fluid collection between the abdominal wall incision and the skin but not draining, Other
Clinical hernia occurrence/recurrence within 12 months after repair. | 12 months
  This study is intended to demonstrate Duramesh superiority to polydioxanone for the development of incisional hernia by 1 year for a laparotomy closure.
Return to the operating room (re-interventions) within 12 months for device related issue. | 12 months
  Re-interventions are defined as: All re-interventions relating to abdominal wall closure complications or abdominal re-exploration.
Surgeon satisfaction at index-procedure using the 5-point smiley face scale. | Procedure
Surgeon satisfaction at 1-month follow-up using the 5-point smiley face scale. | 1 month
Technical success of index-procedure. | Procedure
  Technical success is defined as successful abdominal wall closure without unexpected difficulties.
Device performance using the 5-point smiley face scale. | Procedure
Pain of the surgical incision using 11 point Numeric Pain Rating Scale (NRS) at 1-month follow-up. | 1 month
  The pain NRS is a single 11-point numeric scale with 0 representing one pain extreme (e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable"). The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondents selects a whole number (0 to 10 integers) that best reflects the intensity of their pain. Pain will be scored in rest and with activity. Activity is defined as activity of daily living, e.g. walking, driving, getting into a car, setting the dinner table, doing the laundry, etc.
Pain of the surgical incision using 11 point Numeric Pain Rating Scale (NRS) at 12-months follow-up. | 12 months
  The pain NRS is a single 11-point numeric scale with 0 representing one pain extreme (e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable"). The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondents selects a whole number (0 to 10 integers) that best reflects the intensity of their pain. Pain will be scored in rest and with activity. Activity is defined as activity of daily living, e.g. walking, driving, getting into a car, setting the dinner table, doing the laundry, etc.
Palpability/sensation of suture used for the repair at 12-months follow-up. | 12 months
  Assessment whether the patient can feel the suture.
Quality of life using Short Form 12 (SF-12) health survey at 12-months follow-up. | 12 months
  The SF-12 Health Survey is a 12-item, patient-reported survey of patient health.
Patient satisfaction at 1-month follow-up 5-point smiley face scale. | 1 month
Patient satisfaction at 12-months follow-up 5-point smiley face scale. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Gent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Yes